CLINICAL TRIAL: NCT07254013
Title: Left Bundle Branch Area Pacing (LBBAP) Monitoring Assistant: Evaluation of Portable ECG Solution
Acronym: LBBOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MicroPort CRM (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: WSEN01
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Bradycardia; Left Bundle Branch Area Pacing; Cardiac Resynchronisation Therapy (CRT); ECG
Keywords: LBBAP ECG MONITORING ASSISTANT
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of Smart ECG system in subject with indication for LBBAP (Experimental): Smart ECG system will be used in addition to EP system in subjects with indication for LBBAP
  Interventions: Device: LBBAP implant

INTERVENTIONS:
Device: LBBAP implant — Use of Smart ECG system during the LBB implant

SUMMARY:
To evaluate the capability to monitor LBB success criteria with the use of a Smart ECG system (ECG monitor, 12 leads ECG cable, ECG viewer software ) during a cardiac device implantation involving the placement of a pacing lead in interventricular septum area

DETAILED DESCRIPTION:
The clinical investigation aims to support physicians with a portable and easy to use solution to display ECG and to provide automatic calculation of key ECG indicators (Left Ventricular Activation time (LVAT) and V6-V1 interval) for LBB implantation procedure. This allows physicians to concentrate on lead placement with the benefice from immediate ECG measurements thanks to the automatic software.

The Smart ECG system is class IIA device and it is composed of:

1. CE-marked Smart ECG, Class IIa medical device (rule 10 Annex VIII of MDR)
2. ECG viewer Software (HookUp SmarV2) (providing 12 lead ECG display + automatic interval measurements + shadow plot for QRS visualization) Class IIa medical device (rule 11 Annex VIII of MDR).
3. CE -marked 12 leads ECG cables radiotransparent and defibrillation proof (Class I device)
4. Commercial PC used in combination with the devices under evaluation

The study is a pre-market, non-pivotal study: HookUp Smart V2 software is a non-implantable Class IIA device, with no interaction with the human body and the demonstration of conformity with general safety and performance requirements is based on the results of non-clinical testing methods alone (as article 61(10) from MDR.

ELIGIBILITY:
Inclusion Criteria:

* Subject with indication for LBBAP using an Electrophysiology ECG monitoring system (EP System) as part of pacemaker or CRT-P or CRT-D implant procedure (de novo implant, device revision or upgrade including LOT-CRT)
* Subject signed and dated the ICF

Exclusion Criteria:

* Incapacitated subject or under guardianship
* inability to understand the purpose of the study
* Minor subjects
* Non menopausal women
* Patients implanted with other electrically active non cardiac devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Capability to monitor LBB success criteria with the use of Smart ECG system | baseline/ procedure
  Proportion of investigators providing an overall favorable assessment (assessed "GOOD or ACCEPTABLE") on a four- point scale (GOOD, ACCEPTABLE, POOR, VERY POOR) on the use of Smart ECG system to achieve LBB area pacing.

SECONDARY OUTCOMES:
The accuracy of the two measurements (LVAT and V6-V1) | baseline/ procedure
  The accuracy of the two measurements (LVAT and V6-V1) during the final LBB lead position (LBBAP) will be assessed separately by comparing manual and automatic methods.
Identification of LBB transitions | baseline/ procedure
  Concordance between EP and Smart ECG for the identification of LBB transitions (non-selective to selective or non-selective to LVSP, during threshold test at final lead position)
Type of LBB capture | baseline/ procedure
  Concordance of type of LBB capture as determined by EP vs Smart ECG signals (LBBAP, likely LBBAP, LVSP) - based on centralized blinded review of EP annotated screenshot and Smart ECG recordings
Signal quality analysis | baseline/ procedure
  Comparison of Smart ECG versus EP signal quality analysis (signal to noise ratio, frequency analyses)
Investigator's satisfaction | baseline/ procedure
  Investigator's satisfaction questionnaire about using Smart ECG system during the full procedure (i.e .setting the system for the procedure, monitoring lead progression, assessing pacing capture)
Safety reporting | baseline/ procedure
  To report any SADE, ADE, DD occurred during the investigational procedure

CONTACTS AND LOCATIONS:
Overall Officials: Dr Pierre- Antoine Catalan, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (4):
- France (4):
  - CHU de Besançon, Besançon, France
  - Clermont Ferrand, Clermont-Ferrand, France
  - CHU Grenoble Alpes, Grenoble, France
  - Clinique du Millénaire, Montpellier, France